CLINICAL TRIAL: NCT04481555
Title: Eosinophil-guided Reduction of Inhaled Corticosteroids
Acronym: COPERNICOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COPERNICOS_JUJCPR; 2020-003014-12 (EudraCT Number)
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COPD; Inhaled Corticosteroid; Azithromycin; COPD Exacerbation; Pneumonia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: 4-arm facultative designed, randomized controlled, multicenter, parallel group, double-blinded (azithromycin), non-inferiority intervention study in patients with severe and very severe COPD study.
  Participants will be randomly allocated to one of four treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eosinophil_"Control"/Azithro_"Control" (No Intervention): 1. Azithromycin: patients are given placebo
  2. ICS: The patients are given the usual LAMA/LABA/ICS product in the usual dose.
- Eosinophil_"Active"/Azithro_"Control": (Experimental): a. Azithromycin: placebo b. ICS: All patients will receive LABA/LAMA medication. The ICS medication will be switched on/off according to the most recent blood eosinophil count (at inclusion + every 3 months): i. If blood eosinophil ≥ 300 cells/μL, ICS in usual dose next 3 months. Blood eosinophils are measured every 3 months.
  ii. If blood eosinophil <300 cells/μL, ICS is discontinued.
  Interventions: Drug: ICS
- Eosinophil_"Control"/Azithro_"Active" group (Experimental): Azithromycin: 250 mg azithromycin three times weekly. b. ICS: The patients are given the usual LAMA/LABA/ICS product in the usual dose, where the medical treatment for severe COPD is unchanged throughout the entire project period
  Interventions: Drug: Azithromycin
- Eosinophil_"Active"/Azithro_"Active": (Experimental): 1. Azithromycin: 250 mg azithromycin three times weekly.
  2. ICS: All patients will receive LABA/LAMA medication. The ICS medication will be switched on/off according to the most recent blood eosinophil count (at inclusion + every 3 months):
  Interventions: Drug: Azithromycin; Drug: ICS

INTERVENTIONS:
Drug: Azithromycin — Prophylactic azithromycin treatment 250 mg three times weekly vs placebo
  Arms: Eosinophil_"Active"/Azithro_"Active":; Eosinophil_"Control"/Azithro_"Active" group
Drug: ICS — All patients will receive LABA/LAMA medication. The ICS medication will be switched on/off according to the most recent blood eosinophil count (at inclusion + every 3 months) vs continued LABA/LAMA/ICS treatment
  Arms: Eosinophil_"Active"/Azithro_"Active":; Eosinophil_"Active"/Azithro_"Control":

SUMMARY:
Clinical trial on eosinophil-guided time-updated person-specific reduction of inhaled corticosteroid (ICS) therapy and prophylactic azithromycin therapy in patients with severe or very severe chronic obstructive pulmonary disease (COPD) receiving long-acting b-agonist (LABA) / long-acting muscarinic receptor antagonists (LAMA) / ICS treatment.

DETAILED DESCRIPTION:
Inhaled corticosteroid (ICS) treatment is recommended by Global Initiative for Obstructive Lung Disease (GOLD) for patients with frequent and/or servere exacerbations and blood eosinophils > 0.3 x 10^9 cells/L and in those with ≥ 0,1 x 109 cells blood-eosinophils and recurrent exacerbations while on bronchodilators. ICS treatment, however, is associated with side effects such as diabetes, osteoporosis and pneumonia which is costly for both patients and society. By studying the effects of a personalized, eoseosinophil-guided approach to direct ICS in COPD patients with frequent AECOPDs through a randomized clinical trial this study will examine the possibilities of reducing ICS overtreatment and thus ICS-related adverse events.

Long term ICS treatment is known for affecting the bacterial load in stable COPD patients. Azithromycin exerts multiple effects on the structure and composition of the lower airway microbiota and has anti-inflammatory effects. This study will, moreover, investigate whether an oral low-dose prophylactic treatment with Azithromycin 250 mg three times weekly can reduce the number of moderate-severe AECOPD and improves time alive and out of hospital.

This study is a randomized, double-blinded, multicentre, four-arm intervention clinical trial and is conducted based on the principles of good clinical practise (GCP).

ELIGIBILITY:
Inclusion Criteria:

* COPD (verified by a specialist in respiratory medicine + spirometry)
* GOLD class E anytime within the last 2 years (corresponding to 2 ≥ AECOPD and/or ≥1 AECOPD leading to hospitalization during a 12 months period within the last 2 years) and/or FEV1<30%.
* Treatment for last 4 weeks including LAMA, LABA and ICS
* Informed consent

Exclusion Criteria:

* Known asthma.
* Male < 40 years.
* Female <40 years, if non-menopausal (had menstruation within the last 12 months) conditioned by a negative urine HCG test
* Severe mental illness which considerably complicates co-operation.
* Language problems that considerably complicate co-operation.
* Current treatment with systemic corticosteroids corresponding to > 5 mg prednisolone per day.
* Systemic antibiotic treatment (if to participate in microbiota sub-study) or systemic corticosteroid treatment within 14 days (also prophylactic Azithromycin).
* Contra-indication to treat with Azithromycin (as listed by the producer).
* Non-bacterial exacerbation per investigator judgement in the last 3 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Exacerbations, hospital and death | 365 days
  Number of hospitalization-requiring exacerbations within 12 months and/or death within 365 days

SECONDARY OUTCOMES:
Days alive, out of hospital | 365 days
  Days alive and out of hospital within 365 days after recruitment
Deaths, uncontrolled AECOPD | 365 days
  Death or uncontrolled AECOPD tendency within 365 days
Number of exacerbations | 365 days
  Number of moderate/severe exacerbation within 365 days
Cumulative ICS dose | 365 days
  Cumulative dose of inhaled corticosteroids within 365 days
Cumulative OCS dose | 365 days
  Cumulative dose of systemic corticosteroids within 365 days
Change in FEV1 | 365 days
  Change in lung function (ΔFEV1) from baseline to 365 days
Change in blood eosinophils | 365 days
  Change in blood eosinophils from baseline to 365 days (eosinophilic trajectories)
Diabetes mellitus | 365 days
  New diagnosis of diabetes mellitus within 365 days
Change in HbA1c | 365 days
  Change in HbA1c from baseline to 365 days
Number of antibiotic requiring infections | 365 days
  Antibiotic-requiring infections within 365 days
Microbiota, abundance and diversity | 365 days
  Difference in respiratory microbiota abundance and diversity from baseline to 12 months between treatment arms
Microbiota, immunological profile | 365 days
  Difference in immunological profile including cytokines and chemokines in the upper airways from baseline to 12 months between treatment arms
Change in CAT score | 365 days
  Change in COPD-related quality of life (Based on COPD Assessment Test - CAT) from baseline to 365 days
Change in MRC dyspnoea score | 365 days
  Number who progress to MRC -dyspnea score from < 3 to ≥3 anytime during follow-up (assessed every 3 months).
Number of non-invasive ventilation (NIV) or intensive care admissions or death | 365 days
  Number of admission requiring non-invasive ventilation (NIV) treatment or admissions to intensive care within 365 days
Mortality | 365 days
  Mortality within 365 days

CONTACTS AND LOCATIONS:
Locations (9):
- Denmark (9):
  - Aarhus University Hospital, Aarhus
  - Hvidovre Hospital, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Gentofte Hospital, Hellerup
  - Nordsjællands Hospital, Hillerød
  - Næstved-Slagelse-Ringsted Sygehus, Næstved
  - Odense University Hospital, Odense
  - Roskilde Sygehus, Roskilde
  - Silkeborg Sygehus, Silkeborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ronn C, Bonnesen B, Alispahic IA, Tonnesen LL, Kjaergaard JL, Moberg M, Ulrik CS, Harboe ZB, Browatzki A, Jensen TT, Meyer CN, Bodtger U, Bendstrup E, Johansson SL, Kaiser DU, Hyldgaard C, Vestbo J, Sivapalan P, Jensen JS. Study protocol: COPD-eosinophil-guided reduction of inhaled corticosteroids (COPERNICOS) : A randomized, double-blinded, multicenter, four-arm intervention clinical trial on eosinophil-guided time-updated person-specific reduction of inhaled corticosteroid therapy and prophylactic low dose Azithromycin therapy in patients with severe or very severe chronic obstructive pulmonary disease (COPD). Trials. 2025 Sep 2;26(1):335. doi: 10.1186/s13063-025-09032-0. PMID 40898355